CLINICAL TRIAL: NCT07313683
Title: Lumbopelvic Stabilization Exercises vs. Hypopressive Exercises for Postpartum Recovery: A Randomized Clinical Trial
Brief Title: Therapeutic Exercise for Postpartum Recovery
Acronym: PelviRecover
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alcala (Other)
Responsible Party: Principal Investigator, Virginia Prieto Gómez, Principal Investigator, University of Alcala
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CEIP/2025/3/069
Record Dates: First submitted 2025-11-17; First posted 2026-01-02 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Postpartum Period; Pelvic Floor Disorders
Keywords: Therapeutic exercise; Physical therapy; Intra-abdominal pressure; Pelvic floor; Postpartum period; Quality of life
MeSH Terms: conditions — Pelvic Floor Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The investigator responsible for participant randomization and the statistician performing the data analysis will be masked to group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group 2: Multimodal Physiotherapy (HE + PFMT + TE) (Experimental): Hypopressive Exercises & Pelvic Floor Exercises & Therapeutic Education
  Interventions: Behavioral: Therapeutic Education (TE); Other: Pelvic Floor Exercises (PFMT); Other: Hypopressive Exercises (HE)
- Experimental Group 1: Multimodal Physiotherapy (LSE + PFMT + TE) (Experimental): Lumbopelvic Stabilization Exercises & Pelvic Floor Exercises & Therapeutic Education
  Interventions: Behavioral: Therapeutic Education (TE); Other: Pelvic Floor Exercises (PFMT); Other: Lumbopelvic Stabilization Exercises (LSE)

INTERVENTIONS:
Behavioral: Therapeutic Education (TE) — The participants will receive Therapeutic Education supported by audiovisual materials covering abdominopelvic anatomy and physiology, common dysfunctions, risk factors, and protective strategies, delivered through 4 face-to-face sessions of 20 minutes over the 8-week intervention period.
Other: Pelvic Floor Exercises (PFMT) — The participants will attend 8 weekly 45-minute sessions (4 in person at the Research Group laboratory and 4 online via Physitrack®). They will undergo Pelvic Floor Muscle Training guided intravaginally using manometry biofeedback to improve proprioception, strength, endurance, and relaxation, and will perform the exercises at home at least four times per week.
Other: Lumbopelvic Stabilization Exercises (LSE) — Participants will attend 8 weekly 45-minute sessions (4 in person at the Research Group laboratory and 4 online via Physitrack®). They will perform lumbopelvic stabilization exercises guided by transabdominal ultrasound to ensure correct activation of trunk stabilizing muscles, primarily the transversus abdominis and pelvic floor muscles. Exercises will emphasize coordination of the lumbar multifidus, transversus abdominis, and pelvic floor across different positions, progressing to dynamic tasks involving additional lumbopelvic muscles, light weight lifting, and controlled impact activities such as jump squats. Participants perform the exercises at home at least four times per week.
  Arms: Experimental Group 1: Multimodal Physiotherapy (LSE + PFMT + TE)
Other: Hypopressive Exercises (HE) — Participants will attend 8 weekly 45-minute sessions (4 in person at the Research Group laboratory and 4 online via Physitrack®). They will perform hypopressive exercises under transabdominal ultrasound guidance following the Caufriez method, without voluntary abdominal or pelvic floor contraction, and will perform the exercises at home at least four times per week.
  Arms: Experimental Group 2: Multimodal Physiotherapy (HE + PFMT + TE)

SUMMARY:
Pelvic floor dysfunctions (PFDs) are common conditions that affect women, especially after vaginal childbirth. These disorders can cause urinary or fecal incontinence, pain during sexual activity, and prolapse of pelvic organs, leading to a significant decrease in quality of life. Current scientific evidence shows that early and specific physiotherapy-based interventions after childbirth may help reduce the risk of developing long-term PFDs.

Pelvic floor muscle training (PFMT) is currently the first-line conservative treatment for women with PFD, but in recent years other exercise methods, such as hypopressive exercises, have become increasingly popular, despite limited supporting evidence. At the same time, some women need to return early to physically demanding jobs or impact sports, but there are no clear guidelines on how to safely prepare the abdominopelvic region for progressive exposure to increased intra-abdominal pressure.

This study aims to compare two postpartum recovery exercise programs:

A program based on lumbopelvic stabilization exercises that progressively expose women to increases in intra-abdominal pressure and impact activities.

A program based on hypopressive exercises, which focus on avoiding intra-abdominal pressure.

The goal is to determine which approach is safer and more effective in improving pelvic floor recovery after childbirth and in supporting women in their gradual return to daily, work, and sports activities.

DETAILED DESCRIPTION:
Pelvic floor dysfunctions (PFDs) are highly prevalent conditions that impose a substantial burden on women's health, particularly following vaginal childbirth. Vaginal delivery has been identified as a major risk factor due to potential trauma to the pelvic floor, including overstretching of muscles and nerves, damage to connective tissue supporting pelvic organs, and direct perineal injury. Obstetric interventions such as forceps or vacuum-assisted delivery, episiotomy, and epidural anesthesia may further exacerbate the risk of PFDs. Longitudinal studies indicate that a considerable proportion of women continue to experience urinary or fecal incontinence, dyspareunia, or prolapse for many years after childbirth, highlighting the chronic nature of these dysfunctions and the need for preventive strategies.

Physiotherapy-based interventions have demonstrated promise in reducing the incidence and severity of PFDs when applied early in the postpartum period. Pelvic floor muscle training (PFMT) is considered the gold standard conservative therapy, supported by randomized controlled trials and systematic reviews. PFMT effectively improves muscle strength and function, and its use is endorsed by international guidelines, such as those from the National Institute for Health and Care Excellence (NICE).

In recent years, hypopressive exercises (HE) have been promoted as an alternative or complementary approach to PFMT. HE were originally developed to restore abdominal wall function without provoking increases in intra-abdominal pressure, which is considered a risk factor for pelvic floor overload. Preliminary studies suggest potential benefits in muscle activation and patient satisfaction, yet the quality of evidence remains low, with most research limited to observational designs, small sample sizes, and short follow-up periods. Therefore, the effectiveness and safety of HE in postpartum populations remain uncertain.

Parallel to this, lumbopelvic stabilization exercises (LSE) have been proposed as a means to strengthen the transversus abdominis, multifidus, and pelvic floor muscles through a staged protocol beginning with isometric and coordinated contractions and progressing to integrated functional tasks. Importantly, LSE involve gradual exposure to increased intra-abdominal pressure and impact-related forces, which may facilitate safer return to occupational or athletic activities requiring lifting or high-impact loading. While these exercises have shown benefit in postpartum lumbopelvic pain, there is insufficient evidence on their role in pelvic floor recovery.

Given the growing number of women who resume physically demanding work or impact sports shortly after childbirth, the absence of clear, evidence-based guidelines for abdominopelvic conditioning represents a significant gap in postpartum care. The International Continence Society (ICS) has described PFDs as a "silent epidemic," underlining the urgent need for preventive and rehabilitative interventions supported by rigorous clinical trials.

The present randomized controlled trial is designed to address this gap by directly comparing two structured postpartum rehabilitation approaches: (1) a program of lumbopelvic stabilization exercises incorporating progressive exposure to intra-abdominal pressure and impact, and (2) a program of hypopressive exercises aimed at minimizing intra-abdominal pressure.

This study is expected to generate high-quality evidence regarding the comparative safety and efficacy of these two exercise-based strategies. The findings will provide valuable guidance for clinicians, physiotherapists, and policymakers, contributing to the development of standardized postpartum rehabilitation protocols. Ultimately, the trial seeks to improve long-term pelvic health outcomes and support women in safely returning to their daily, occupational, and athletic activities after childbirth.

ELIGIBILITY:
Inclusion Criteria

* Primiparous or multiparous women with an uncomplicated vaginal delivery.
* Women between 6 and 12 weeks postpartum.
* Women who have freely read, understood, and signed the informed consent form.

Exclusion Criteria

* Cesarean delivery.
* Pelvic or perineal pain greater than 4/10 during physical examination.
* Clinical diagnosis of pelvic floor myofascial pain syndrome.
* Evidence of levator ani muscle avulsion.
* Third- or fourth-degree perineal tears.
* History of pelvic surgery.
* History of pelvic fractures and/or pelvic neoplasms.
* Current pregnancy.
* Neurological disorders.
* Active vaginal or urinary tract infections.
* Cognitive, auditory, or visual impairments that limit comprehension, questionnaire completion, consent, or participation in the study.
* Individuals under 18 years of age.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Only individuals whose biological sex is female are eligible to participate, as the study involves postpartum women. Eligibility is based on having experienced childbirth, regardless of gender identity.
Enrollment: 84 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2028-09 (Estimated); Study Completion 2029-01 (Estimated)

PRIMARY OUTCOMES:
Health-related quality of life (HRQoL) | Baseline (V0); immediately after completing the intervention (V1); 3 months (V2); 6 months (V3); and 12 months (V4) after intervention.
  Self-administration of the PFDI-20 questionnaire, which evaluates urogenital, anorectal, and prolapse-related symptoms. Each subscale ranges from 0 to 100, with lower scores indicating better quality of life (less symptom distress).

SECONDARY OUTCOMES:
Sexual function | Baseline (V0); immediately after completing the intervention (V1); 3 months (V2); 6 months (V3); and 12 months (V4) after intervention.
  Self-administration of the Female Sexual Function Index (FSFI), which assesses sexual function across six domains: desire, arousal, lubrication, orgasm, satisfaction, and pain. The FSFI total score ranges from 2 to 36. A cutoff score of <27 is commonly used to indicate sexual dysfunction
Physical activity level | Baseline (V0); immediately after completing the intervention (V1); 3 months (V2); 6 months (V3); and 12 months (V4) after intervention.
  Self-administration of the International Physical Activity Questionnaire (IPAQ). This instrument estimates weekly physical activity based on energy expenditure expressed in MET·min/week, taking into account the frequency, duration, and intensity of the activities performed. It classifies individuals into three categories: low (inactive), moderate, or high.
Urogenital hiatus distance | Baseline (V0); immediately after completing the intervention (V1); 3 months (V2); 6 months (V3); and 12 months (V4) after intervention.
  2D transperineal ultrasound (Mindray M7, Shenzhen, China): sagittal plane, measuring the distance between the inferior margin of the pubic symphysis and the anorectal angle. Measurements will be obtained at rest and during maximal pelvic floor muscle contraction.
Pelvic floor muscle tone and strength | Baseline (V0); immediately after completing the intervention (V1); 3 months (V2); 6 months (V3); and 12 months (V4) after intervention.
  Vaginal dynamometry (Pelvimetre, Phenix Vivaltis, Montpellier, France): in the lithotomy position, resting tone will be recorded as the lowest value obtained with the pelvic floor muscles relaxed, and strength will be determined as the mean of three maximal voluntary contractions.
Perceived self-efficacy | Baseline (V0); immediately after completing the intervention (V1); 3 months (V2); 6 months (V3); and 12 months (V4) after intervention.
  Self-administration of the Broome Pelvic Muscle Self-Efficacy Scale: this instrument evaluates self-efficacy expectations regarding the performance of specific pelvic floor muscle exercises and the anticipated outcomes. The maximum score is 100, indicating high self-efficacy, while scores below 33 reflect low self-efficacy.
Functional capacity | Baseline (V0); immediately after completing the intervention (V1); 3 months (V2); 6 months (V3); and 12 months (V4) after intervention.
  30-Second Sit-to-Stand Test: records the total number of complete repetitions of standing up from and sitting down on a standard armless chair, with the arms crossed over the chest, performed within a 30-second interval.

OTHER OUTCOMES:
Treatment safety | After each weekly session during the 8-week intervention (Weeks 1-8); immediately post-intervention (V1, Week 8); 3 months (V2), 6 months (V3), and 12 months (V4) post-intervention.
  All adverse events occurring during the intervention period will be recorded, including the onset of pain, medical consultations related to the treatment, medication use, postponement of sessions due to treatment-related issues, or withdrawal from the intervention.
Satisfaction level | Immediately after completing the intervention (V1)
  Verbal numerical scale ranging from 0 to 10, where 0 indicates complete dissatisfaction with the treatment and 10 represents excellent satisfaction.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Nursing and Physiotherapy, University of Alcalá, Alcalá de Henares, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be made available due to privacy and ethical restrictions. Aggregated study results will be published in peer-reviewed journals and may be shared upon reasonable request.